CLINICAL TRIAL: NCT03775408
Title: Femoral Antegrade Starting Tool (FAST): Clinical Feasibility Pilot Study
Brief Title: FAST: Clinical Feasibility
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: FAST2019
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FAST Patients: Patients at Sunnybrook Health Sciences Centre with femur fractures that will undergo a femoral antegrade intramedullary nailing procedure.
  Interventions: Device: FAST

INTERVENTIONS:
Device: FAST — Orthopaedic surgeons will use the FAST device to facilitate entry point selection and alignment of a guidewire for intramedullary nailing of femoral shaft fractures.

SUMMARY:
This study evaluates the clinical ease of use of the Femoral Antegrade Starting Tool (FAST).

DETAILED DESCRIPTION:
The investigators will recruit 10 patients at Sunnybrook Health Sciences Centre that are scheduled to receive femoral antegrade intramedullary nailing to treat a femur fracture. This study evaluates the clinical ease of use of the Femoral Antegrade Starting Tool (FAST) device, and the surgical workflow during entry point selection and guidewire alignment for intramedullary nailing of femoral fractures. It is hypothesized that the usage of the tool will reduce surgery time and number of images required.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a femoral shaft fracture
* Undergoing anterograde intramedullary nailing procedure

Exclusion Criteria:

* Femoral head or neck fractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at Sunnybrook Health Sciences Centre
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure Time | 1 day
  Time of the procedure from the initiation of the guidewire step (surgeon picking up the guidewire) to the removal of the FAST device following acceptable guidewire placement

SECONDARY OUTCOMES:
Fluoroscopic Images | 1 day
  Number of fluoroscopic images used to obtain start point
Number of guidewire drilling attempts | 1 day
  Number of times the guidewire has been drilled into the bone to test the alignment.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Tomescu, MD MSc FRCS, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebrahimi H, Yee A, Whyne C. Surgical process analysis identifies lack of connectivity between sequential fluoroscopic 2D alignment as a critical impediment in femoral intramedullary nailing. Int J Comput Assist Radiol Surg. 2016 Feb;11(2):297-305. doi: 10.1007/s11548-015-1262-6. Epub 2015 Jul 21. PMID 26194487